CLINICAL TRIAL: NCT01427517
Title: Intravenous N-acetylcysteine for the Treatment of Gaucher's Disease and Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWA00000312-2; U54NS065768 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease; Gaucher's Disease
Keywords: Parkinson's disease; Gaucher's disease; Control
MeSH Terms: conditions — Parkinson Disease; Gaucher Disease | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NAC in PD (Experimental): single intravenous administration of N-acetylcysteine in PD patients
  Interventions: Drug: N-acetylcysteine
- NAC in GD (Experimental): single intravenous administration of N-acetylcysteine in GD patients
  Interventions: Drug: N-acetylcysteine
- NAC in controls (Experimental): single intravenous administration of N-acetylcysteine in control subjects
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — Single, intravenous administration of N-acetylcysteine
  Other Names: NAC

SUMMARY:
The investigators are interested in determining if the investigators are able to detect changes in brain chemistry using Magnetic Resonance Spectroscopy (MRS) in individuals with Parkinson's disease (PD), those with Gaucher's disease (GD), and those without neurological disorders (healthy controls) when they are given the antioxidant N-acetylcysteine (NAC). This study will combine information from a medical history, a physical examination and disease rating scales with results obtained using MRS brain scans and pharmacokinetic studies from blood samples. This research will require 1 visit that will require about 4 to 5 hours of time. During this study, participants will provide their medical history, be examined and undergo a rating scale for about one hour; the brain scan and pharmacokinetic studies will require 1.5-2 hours of time; in total the study will take about 4-5 hours.

DETAILED DESCRIPTION:
Oxidative stress is implicated in the pathogenesis of a number of neurodegenerative diseases such as Parkinson's disease (PD). Further, levels of glutathione (GSH), a prevalent endogenous antioxidant, are decreased in the postmortem substantia nigra (SN) of individuals with PD, indicating increased oxidative stress, although this has yet not been confirmed in vivo. Increases in intracellular oxidative stress have also been observed in primary fibroblast cultures obtained from patients with GD, where enzyme replacement therapy resulted in increases in total GSH. The hypothesis that oxidative stress plays a key role in the neurodegeneration associated with PD suggests that antioxidants may be useful in altering disease progression.

N-acetylcysteine (NAC) is a well-known antioxidant that is thought to act both as a free radical scavenger and as a cysteine donor for the synthesis of GSH. NAC may be beneficial in the treatment of PD and GD. Magnetic resonance spectroscopy (MRS) methods may be able to determine if there are effects from NAC on central nervous system GSH levels. In addition, use of red blood cell (RBC) measurements of GSH, if correlated with brain concentrations, could serve as an easily measured biomarker to help characterize and monitor response to therapy. The investigators therefore propose to conduct a study of the effect of a single, intravenous dose of NAC on central (brain) measures of GSH and peripheral (RBC) measures of GSH in people with PD and healthy controls, through the use of simultaneous MRS techniques and pharmacokinetic studies. The investigators hypothesis and specific aims are as follows:

Hypothesis: RBC and brain GSH concentrations will increase following oral NAC administration in individuals with Parkinson's disease (PD), Gaucher's disease (GD), and control participants.

Specific Aims:

1. Quantitate baseline plasma and red blood cell GSH concentrations in those with PD and GD and controls; and characterize NAC and GSH pharmacokinetics after a single intravenous NAC administration.
2. Quantitate brain GSH levels (as ascertained through MRS) in those with PD and GD and controls at baseline and after a single intravenous NAC administration simultaneously with Aim 1.
3. Construct a pharmacokinetic model to evaluate the relationship between peripheral (plasma and RBC) and central (brain) GSH measurements.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must be 18 years or older.
2. All enrollees must understand and cooperate with requirements of the study in the opinion of the investigators and must be able to provide written informed consent.
3. Individuals with medically stable Parkinson's disease (in the opinion of the investigator).
4. All participants must not have taken antioxidants coenzyme Q-10, vitamin C, or vitamin E for 3 weeks prior to the study.
5. Absence of dementia in all subjects, as determined by pre-scanning cognitive assessment.
6. Control subjects who are able to undergo MRS

Exclusion Criteria:

1. Inability to undergo MRI scanning without sedation
2. Medically unstable conditions in any group as determined by the investigators
3. Pregnant or lactating or those women of child-bearing age that are not using acceptable forms of contraception
4. Diagnosis of asthma that is presently being treated with ANY medication, or past history of asthma/bronchospasm resulting in an emergency room visit, hospitalization or treatment
5. Unable to adhere to study protocol for whatever reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tuite, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Holmay MJ, Terpstra M, Coles LD, Mishra U, Ahlskog M, Oz G, Cloyd JC, Tuite PJ. N-Acetylcysteine boosts brain and blood glutathione in Gaucher and Parkinson diseases. Clin Neuropharmacol. 2013 Jul-Aug;36(4):103-6. doi: 10.1097/WNF.0b013e31829ae713. PMID 23860343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were primarily recruited from the investigators' clinics at the University of Minnesota, and from research volunteers signed up with the University's Center for Magnetic Resonance Research.
Pre-assignment Details: Groups were not assigned in this study. All subjects received the same intervention.
Period: Overall Study
Arm/Group | NAC in PD | NAC in GD | NAC in Controls
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAC in PD | NAC in GD | NAC in Controls | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 3 | 2 | 3 | 8
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.33 (3.21) | 44 (23.58) | 58 (0) | 52.11 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 5
  Male | 0 | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Brain GSH
Description: change in brain GSH levels from baseline to post-NAC administration (90 - 110 minutes) in all subjects
Time Frame: Baseline and up to 110 minutes post-NAC administration
Measure: Mean (Standard Deviation); unit: percent increase from baseline
Arm/Group | NAC in PD | NAC in GD | NAC in Controls
Number analyzed (Participants) | 3 | 3 | 3
percent increase from baseline | 55 (24.4) | 41 (16.3) | 34 (19.8)

ADVERSE EVENTS:
Arm/Group | NAC in PD | NAC in GD | NAC in Controls
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC in PD (N=3) | NAC in GD (N=3) | NAC in Controls (N=3)
allergic reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Following scan, a subject complained of itchy of hands, nasal congestion, sore throat. Study staff noted swelling around eyes and flushed cheeks & neck. Subject was taken to ER (not admitted)& received standard treatment for allergic reaction to NAC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes